CLINICAL TRIAL: NCT00576394
Title: Impact of Aggressive Versus Moderate Glycemic Control on Clinical Outcomes Following Coronary Artery Bypass Graft Surgery in Diabetic Patients
Brief Title: Aggressive Versus Moderate Glycemic Control in Diabetic Coronary Bypass Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Heart Association (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Harold L. Lazar MD, Professor of Cardiothoracic Surgery, American Heart Association
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-25760
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Glycemic Control
Keywords: Glucose, Insulin
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1Moderate Glycemic Control (Active Comparator): Patients will receive an insulin drip to keep blood glucose levels between 120-180mg/dl
  Interventions: Drug: IV Insulin drip
- 2Aggressive Glycemic Control (Active Comparator): Patients will receive an insulin drip designed to maintain serum glucose between 80-120mg/dl
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: IV Insulin drip — IV insulin drip at 100units insulin in 100ml saline designed to keep blood glucose between 120-180mg/dl
  Arms: 1Moderate Glycemic Control
Drug: Insulin — IV insulin drip to keep serum glucose between 80-120mg/dl.
  Arms: 2Aggressive Glycemic Control

SUMMARY:
entGlycemic control has been found to improve clinical outcomes following Coronary Bypass Surgery. This study tests the hypothesis that obtaining tighter glycemic control(80-120mg/dl) as opposed to more moderate control (120-180mg/dl) will further improve outcomes.

DETAILED DESCRIPTION:
150 diabetic patients will be randomized to achieve aggressive glycemic control (80-120mg/dl) vs moderate control (120-180mg/dl) using intravenous insulin infusions beginning at anesthetic induction and continuing for 18 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* All diabetic patients undergoing Coronary Bypass Surgery

Exclusion Criteria:

* Patients with hepatic and renal failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2006-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypoglycemia | 24 hours following surgery

SECONDARY OUTCOMES:
free fatty acid levels | 24 hours following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Lazar HL, McDonnell MM, Chipkin S, Fitzgerald C, Bliss C, Cabral H. Effects of aggressive versus moderate glycemic control on clinical outcomes in diabetic coronary artery bypass graft patients. Ann Surg. 2011 Sep;254(3):458-63; discussion 463-4. doi: 10.1097/SLA.0b013e31822c5d78. PMID 21865944